CLINICAL TRIAL: NCT03932539
Title: New Strategies to Improve Immunosuppressive Therapy Management in Heart Transplantation: a Pilot Study
Brief Title: Improving Immunosuppressive Therapy in Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Mariadelfina Molinaro, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 15547/2019
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Rejection Heart Transplant; Immunosuppression
Keywords: Immunosuppressive therapy; Tacrolimus; Heart transplantation; Pharmacokinetics; Pharmacogenetics; Acute rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Twenty-five de-novo heart transplant recipients: Twenty-five de-novo heart transplant recipients will be enrolled, male and female, aging 18-70 years, receiving TAC in combination with steroids and antiproliferative drugs, either Everolimus or Sirolimus.

SUMMARY:
Cardiac allograft rejection (CAR) occurs in 30% to 40% of transplant recipients within the first year post-transplant, and carries an increased risk of both acute graft failure and reduced graft longevity. Because of the high morbidity of CAR when diagnosed after symptoms develop, surveillance endomyocardial biopsy (EMB) has been included in heart transplantation guidelines since 1990. Although EMB is the established gold standard for the diagnosis of CAR, the clinical utility of EMB using standard hematoxylin and eosin (H&E) histologic analysis is limited by marked inter-observer variability and significant discordance between the histologic grade and clinical impression of CAR severity.

On the other hand, Tacrolimus (TAC), one of the most important immunosuppressant drug and widely used for the prevention of rejection after solid organ transplantation (SOT), is considered a critical dose drug: too low exposure to TAC may result in under-immunosuppression and acute rejection, whereas overexposure puts patients at risk for toxicity. Tac concentrations, in whole-blood, are considered therapeutic when maintained in the range 5 and 20 ng/mL. In addition to being highly variable inter-individually, TAC pharmacokinetics can also be variable within individual patients.

Although in recent years significant decrease of rejection post SOT has been observed, there is space for further modulation of immunosuppressive therapy, in order to reduce the most common adverse side effects (nephrotoxicity, diabetes, osteoporosis, cardiovascular disease, infections and malignancies), to improve the patients quality of life and to better individualize their therapies. Tac. Unfortunately, a clear correlation between TAC whole blood concentration and acute rejection risk has not yet been defined.

DETAILED DESCRIPTION:
Monocentric and Observational Study

- Longitudinal Prospective

The study considers the collection of the following samples:

* a single whole blood sample, 3-5 mL in EDTA for Pharmacogenetics,
* 10 mL whole blood sample in lithium-heparin for Tac quantification in PBMC collected at each time-point scheduled for routine follow-up visits: day +15 and month 1, 3, 6, 12 post transplant
* About 1 mg cardiac tissue samples (from cardiac biopsies), collected by standard procedure adopted at the Transplant Center of CardiacSurgery at each time-point scheduled for routine follow-up visits: day +15 and month 1, 3, 6, 12 post transplant

Each blood sample and biopsy specimen will be identified and labeled with an alphanumeric code, whose decoding matrix will be kept by dedicated personnel at the U.O.C. Cardiac Surgery, Department of Intensive Medicine.

In general, each patient will be defined as "TAC + progressive enrollment number" (example: TAC1, TAC2, TAC3 ...).

Each sample sent to the laboratories for the analyzes in the different matrices and for the different activities foreseen by the protocol (measurements of tacrolimus and pharmacogenetic concentrations) must always contain the identification code assigned to the patient followed by the type of analysis + sampling time. For example, patient collection # 2 for tacrolimus assay to be performed in PBMC, whole blood and EMB at month 3, will be identified as:

TAC2-PBMC-M3 TAC2-WB-M3 TAC2-BEM-M3

The storage of the codes that will allow the patients' identification will be kept by dr. Carlo Pellegrini and dr. Barbara Cattadori (U.O.C. Cardiosurgery).

All samples will be investigated within the Foundation: blood samples for the quantification of Tacrolimus in blood mononuclear cells (PBMC) and in whole blood will be transferred to the Clinical and Experimental Pharmacokinetic Laboratory. Blood samples for pharmacogenetic investigations will be transferred to the Biochemical and Genetic Laboratory of Respiratory Diseases.

The proponents of the study will keep any residual samples at the investigations planned by the study in a safe place with limited access, ie in a freezer -80 °C located in a locked room (room n.11a, Lab Clinical and Experimental Pharmacokinetics, Pavilion 13). These samples can be used for scientific purposes directly related to those of the main study

ELIGIBILITY:
Inclusion Criteria:

* de-novo heart transplant recipients
* Male and female (18-70 years)
* Receiving TAC in combination with steroids, antiproliferative drugs, Everolimus, Sirolimus.

Exclusion Criteria:

* Age < 18 years
* Intolerance of the drug object of the present study (Tacrolimus) or at any of the excipients contained therein
* Intolerance to glucose
* Diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: If no contraindications will be observed, and the patient will be able to tolerate the administration of the study drug, the patients will be enrolled within the 5th post-transplant day.
  In the case of impossibility to administer the drug within that period, the patient will not have access to the study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
TAC concentration in whole blood | 2 years
  To detect if a correlation exists between the concentration of tacrolimus in whole blood and the acute transplanted heart rejection.
  TAC concentration in whole-blood samples will be measured in ng/mL
TAC concentration in peripheral blood mononuclear cell (PBMC) | 2 years
  To detect if a correlation exists between the concentration of tacrolimus in PBMC and the acute transplanted heart rejection.
  TAC concentration will be measured in PBMC (pg/million of cells)
TAC concentration in endomyocardial biopsy (EMB) | 2 years
  To detect if a correlation exists between the concentration of tacrolimus in EMB and the acute transplanted heart rejection.
  TAC concentration will be measured in pg/mg of biopsy

SECONDARY OUTCOMES:
Pharmacogenetic analysis | 2 years
  Different single nucleotide polymorphisms (SNPs) will be analyzed in ABCB1 (P-gp) and CYP3A4/CYP3A5 genes

CONTACTS AND LOCATIONS:
Overall Officials: Mariadelfina Molinaro, MScBiol, Principal Investigator — IRCCS Policlinico San Matteo
Locations (4):
- Italy (4):
  - Clinical and Experimental Pharmacokinetics Unit, Pavia
  - Clinical Epidemiology and Biometry Unit, Pavia
  - Department of Cardiac Surgery, Pavia
  - Department of Respiratory Diseases - Biochemical and Genetics Lab., Pavia